CLINICAL TRIAL: NCT01188330
Title: Randomized Study Comparing the Interest of a Program of Evaluation and Geriatric Intervention on the Functional Status, Quality of the Life, and Survival of Elderly Patients With Acute Myeloid Leukaemia. MLSP/IPC 2009-003
Brief Title: Program of Evaluation and Geriatric Intervention on the Functional Status, Quality of the Life, and Survival
Acronym: MLSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MLSP/IPC 2009-003
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Geriatric Assessment; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WITH Comprehensive Geriatric assessment (Experimental): Conventional haematological management of patients and Comprehensive Geriatric assessment (CGA) at diagnosis followed by interventions according to disabilities detected and planned monthly follow up by a nurse practitioner during 6 months.
  Interventions: Behavioral: WITH Comprehensive Geriatric assessment
- Conventional (Active Comparator): Conventional haematological management of patients
  Interventions: Behavioral: Conventional

INTERVENTIONS:
Behavioral: WITH Comprehensive Geriatric assessment — Each month after randomization, a nurse practitioner will systematically review the intervention plan.
  In case of hospitalisation, the nurse will go and meet the patient and his care giver to check each point of the intervention plan. If an action has not been done, a new proposal will be made to the patient. If the patient is at home or in institution, the nurse practitioner will call the patient and /or his care giver for the same purpose
  Arms: WITH Comprehensive Geriatric assessment
Behavioral: Conventional — no Comprehensive Geriatric assessment
  Arms: Conventional

SUMMARY:
Acute myeloid leukaemia (AML) is a disease of the elderly, with a median age at diagnosis of 65. A poor outcome in this population has been well established, with very short overall survival (OS) and disease free survival (DFS).There are numerous bad prognostic factors related to the disease itself or to the patient's medical condition.

This study will evaluate the impact of a Comprehensive Geriatric assessment (CGA) performed at diagnosis with planned interventions according to disabilities and monthly follow-up by a nurse practitioner during 6 months on functional status of older cancer patients treated for Acute myeloid leukaemia. Functional status will be assessed with the Lawson Instrumental Activities of Daily Living (IADL) scale at diagnosis and 6 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years and older
* Referred for treatment following a diagnosis of acute myeloid leukaemia.
* signed informed consent

Exclusion Criteria:

* Terminal patients, with a life expectancy estimated to be less than 3 months, will be excluded from the study, due to ethical issues and the fact that they are unlikely to benefit from this evaluation.
* Patients unable to give informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
functional status | 6 months
  The functional status is evaluated with KATZ INDEX : BASIC ACTIVITIES OF DAILY LIVING (ADL) and Older American Resources and Services, Instrumental Activities of Daily Living (IADL) mesured at diagnosis and 6 month after inclusion.

SECONDARY OUTCOMES:
nutritional status | 6 months
  mesured by the Mini Nutritional Assessment Short Form (mini MNA-SF)
quality of life | 6 months
  estimated by a Quality of Life Questionnaire including 30 items (QLQ-C30)
survival | 6 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Aude CHARBONNIER, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Aude CHARBONNIER, MD, Marseille
  - Christian RECHER, Toulouse

REFERENCES:
- See also: institut Paoli-Calmettes web site — http://www.institutpaolicalmettes.fr/